CLINICAL TRIAL: NCT01783080
Title: Behavioral Activation (BA) for Medication-responsive Chronically Depressed Patients With Impaired Social Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #5908
Record Dates: First submitted 2013-01-25; First posted 2013-02-04 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-04

CONDITIONS: Persistent Depressive Disorder
Keywords: Chronic depression; Dysthymic disorder; Double Depression; Behavioral Activation therapy; Work impairment; Unemployment
MeSH Terms: conditions — Dysthymic Disorder | interventions — Return to Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral Activation for Return to Work (Experimental): BA is a manualized psychotherapy with comparable efficacy to cognitive behavioral treatment and antidepressant medication for acute treatment of depression. In this study, BA's focus was shifted to target work dysfunction by activating the patient into employment-related goals. BA-W consisted of 12 50-minute weekly sessions. Conceptualizing work dysfunction as a product of avoidance patterns and low levels of positive reinforcement, the treatment addressed maladaptive coping strategies such as avoidance as maintaining work dysfunction beyond remission of symptoms. Rather than broadly activating patients, activity scheduling focused on tasks such as sending out resumes, calling for job interviews, and networking to meet potential employers.
  Interventions: Behavioral: Behavioral Activation for return to work

INTERVENTIONS:
Behavioral: Behavioral Activation for return to work — See Arm Description

SUMMARY:
The investigators aimed to assess the ability of a modified version of Behavioral Activation for occupational and social improvement to produce change in: 1. social adjustment, 2. work functioning, 3. avoidance behavior and 4. behavioral activation.

DETAILED DESCRIPTION:
Psychosocial functioning was assessed before and after BA treatment in medication responsive depressed individuals who continued to have impaired social functioning. The primary goal was to demonstrate feasibility of recruitment and retention, and obtain an open pilot sense as to whether there are benefits from this brief psychotherapy approach in this population. The investigators also planned to refine measures and estimate the effect size of any treatment response to estimate power and sample size with the goal of completing a future controlled study.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20-75 years
* a primary diagnosis of Dysthymic Disorder, Chronic major depressive disorder or double depression
* a >50% decrease in 17 item Hamilton Rating Scale for Depression (HRSD-17) score and a final HRSD-17 score ≤ 10 with an adequate antidepressant medication (ADM) trial (> 4 weeks on at least 50% Physician's Desk Reference maximum ADM dose)
* a rating of 1 ("very much improved") or 2 ("much improved") on the Clinical Global Impressions-Improvement scale (CGI-I)
* continued functional impairment, defined by scores >1.9 on the Social Adjustment Scale (SAS)
* unemployment (jobless, looking for work) according to the Bureau of Labor Statistics: jobless and looking and available for work, or underemployed.

Exclusion Criteria:

* Structured Clinical Interview for Diagnostic and Statistical Manual, fourth edition (DSM-IV) Axis I disorders-diagnosed cognitive or psychotic disorders
* bipolar disorder
* active eating disorders
* severe borderline personality disorder
* alcohol or drug dependence (except nicotine) in the last 6 months
* current suicide risk
* unstable medical conditions
* use of psychotropic medications other than antidepressants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Hellerstein, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson G, Hellerstein DJ. Behavioral activation therapy for remediating persistent social deficits in medication-responsive chronic depression. J Psychiatr Pract. 2011 May;17(3):161-9. doi: 10.1097/01.pra.0000398409.21374.ab. PMID 21586994
- [Result] Hellerstein DJ, Erickson G, Stewart JW, McGrath PJ, Hunnicutt-Ferguson K, Reynolds SK, O'Shea D, Chen Y, Withers A, Wang Y. Behavioral activation therapy for return to work in medication-responsive chronic depression with persistent psychosocial dysfunction. Compr Psychiatry. 2015 Feb;57:140-7. doi: 10.1016/j.comppsych.2014.10.015. Epub 2014 Nov 7. PMID 25464836

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation for Return to Work: BA is a manualized psychotherapy with comparable efficacy to cognitive behavioral treatment and antidepressant medication for acute treatment of depression. BA has two primary foci: 1) functional analyses of cognitive and behavioral processes that involve avoidance and 2) using avoided activities to guide activity scheduling. In this study, BA's focus was shifted to target work dysfunction by activating the patient into employment-related goals. BA-W consisted of 12 50-minute weekly sessions. Conceptualizing work dysfunction as a product of avoidance patterns and low levels of positive reinforcement, the treatment addressed maladaptive coping strategies such as avoidance as maintaining work dysfunction beyond remission of symptoms. Rather than broadly activating patients, activity scheduling focused on tasks such as sending out resumes, calling for job interviews, and networking to meet potential employers.
  Behavioral Activation for return to work: See Arm Description
Period: Overall Study
Arm/Group | Behavioral Activation for Return to Work
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Activation for Return to Work
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Paid Work Hours at Week 12
Description: Subject-reported paid work hours per week at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Behavioral Activation for Return to Work
Number analyzed (Participants) | 16
hours | 30.3 (18.8)
Statistical Analysis 1: Comparison: Behavioral Activation for Return to Work; Test type: Superiority or Other; p = 0.005, Regression, Linear; Mean Difference (Final Values) = 13.4

2. Primary Outcome: Paid Work Hours at Week Baseline
Description: Subject-reported paid work hours per week at week baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Behavioral Activation for Return to Work
Number analyzed (Participants) | 16
hours | 16.9 (16.2)

3. Secondary Outcome: Social Functioning at Week Baseline on the Social Adjustment Scale
Description: Social adjustment was measured using the Social Adjustment Scale (SAS). The SAS is a self-report scale that assesses depressive symptoms and functioning in nine social and work-related domains generating a total score that is indicative of a subject's overall level of social adjustment. Subjects rate their own social functioning over times on a 5-point scale on items covering work for pay, housework, extended family, parenting, marital status, social activity and leisure, family unit and student status (sub-scales). Mean values of all the sub-scales are used, with a range from 0-5. Higher score = worse outcome … worse functioning
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: unites on a scale
Arm/Group | Behavioral Activation for Return to Work
Number analyzed (Participants) | 16
unites on a scale | 2.4 (0.5)
Statistical Analysis 1: Comparison: Behavioral Activation for Return to Work; Test type: Superiority or Other; p = 0.11, Regression, Linear; Mean Difference (Final Values) = -0.26

4. Secondary Outcome: Social Functioning at Week 12 on the Social Adjustment Scale
Description: as for outcome 3
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: unites on a scale
Arm/Group | Behavioral Activation for Return to Work
Number analyzed (Participants) | 16
unites on a scale | 2.18 (0.6)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Behavioral Activation for Return to Work
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
This was a small open treatment study, without a comparator group and with limited followup. Findings of this pilot study should be replicated in a larger prospective trial with a randomized design, and with longer followup.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No